CLINICAL TRIAL: NCT01775553
Title: Recapturing Disease Response: A Phase II Study of High Dose Carfilzomib in Patients With Relapsed or Refractory Multiple Myeloma Who Have Progressed on Standard Dose Carfilzomib
Brief Title: Study of High Dose Carfilzomib in Multiple Myeloma Patients Who Have Progressed On Standard Dose Carfilzomib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ajai Chari (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Ajai Chari, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-1506; CAR IST 534
Record Dates: First submitted 2012-09-25; First posted 2013-01-25 (Estimated); Results first posted 2017-06-21 (Actual); Last update posted 2017-06-21 (Actual); Status verified 2017-05

CONDITIONS: Relapse Multiple Myeloma; Refractory Multiple Myeloma
Keywords: Relapsed Multiple Myeloma; Refractory Multiple Myeloma; High-Dose Carfilzomib; Standard Dose Carfilzomib; Carfilzomib
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Carfilzomib (Experimental): All patients will receive Carfilzomib
  Interventions: Drug: Carfilzomib

INTERVENTIONS:
Drug: Carfilzomib — During Cycle 1, patients will receive either 20 mg/m2 on days 1,2 (if the subject has not received carfilzomib as part another clinical trial within the last 4 weeks) or 56 mg/m2 (if the subject is enrolling in the present study after progression of disease on carfilzomib within the last month - for example subjects enrolled in CMAP compassionate use carfilzomib). Thereafter, all subjects will receive 56 mg/m2 for the remaining doses given Cycle 1 Day 8 onwards. Each cycle is 28 days.
  Other Names: High Dose Carfilzomib

SUMMARY:
The purpose of this study is to determine the safety and activity of the investigational drug known as carfilzomib in the treatment of multiple myeloma (MM) when it is given at doses above the usual dose after the standard dosing has become ineffective. The other purpose of this study is to understand what causes the multiple myeloma to become resistant to carfilzomib and whether this can be overcome in the laboratory.

DETAILED DESCRIPTION:
This is an open label, single center, phase II study of high dose carfilzomib. Patients with relapsed or relapsed/refractory myeloma and with progression of disease on standard dosing (20/27 mg/m2) and schedule of carfilzomib will be initially treated at dose level 1, carfilzomib 20/56 mg/m2. During Cycle 1, patients will receive either 20 mg/m2 on days 1,2 (if the subject has not received carfilzomib as part another clinical trial within the last 4 weeks) or 56 mg/m2 (if the subject is enrolling in the present study after progression of disease on carfilzomib within the last month - for example subjects enrolled in CMAP compassionate use carfilzomib). Thereafter, all subjects will receive 56 mg/m2 for the remaining doses given Cycle 1 Day 8 onwards. If a minimal response or better is achieved (and therefore disease response is recaptured) a bone marrow biopsy will be repeated.

If 56 mg/m2 is not tolerated, the dose of carfilzomib will be reduced to dose level -1 i.e. 45 mg/m2. If a subject does not tolerate 45 mg/m2 then the dose would be further reduced to dose level -2 i.e. 36 mg/m2. If the subject does not tolerate 36 mg/m2, then this subject would have to come off study.

Dexamethasone 8 mg po/IV will be administered prior to all carfilzomib doses.

Once a patient develops disease progression on this study, the patient may return to receiving the maximum tolerated dose of carfilzomib by that patient with the addition of a therapeutic dosing of dexamethasone (a total of 20-40 mg weekly). An IMId (e.g. thalidomide or lenalidomide) and/or an alkylator can also be added to carfilzomib 27 or 36 mg/m2 per investigator discretion either concurrent with the addition of dexamethasone or subsequent to disease progression on carfilzomib with concurrent therapeutic dexamethasone.

ELIGIBILITY:
Inclusion Criteria:

Disease-related:

1. Multiple myeloma
2. Subjects must have measurable disease, defined as one or both of the following:

   1. Serum M-protein ≥ 1.0 g/dL
   2. Urine M-protein ≥ 200 mg/24 hours
   3. Free light chains: Only in patients without measureable serum and urine M-protein levels: the difference between involved and uninvolved FLC levels must be at least 10 mg/dl.
3. Refractory to the most recently received therapy. Refractory disease is defined as ≤ 25% response or progression during therapy or within 60 days after completion of therapy.
4. Subjects must have progressed on standard dose 20/27 mg/m2 and schedule of carfilzomib without having had any carfilzomib related grade 3 or 4 toxicities.
5. Subjects must have received ≥ 2 prior regimens for relapsed disease. Induction therapy and stem cell transplant will be considered as one regimen
6. Subjects must have received prior treatment with bortezomib, and either thalidomide or lenalidomide
7. Subjects must have received an alkylating agent unless contraindicated. Subjects may have received these agents alone or in combination with other myeloma treatments.

Demographic:

1. Age ≥ 18 years
2. Life expectancy ≥ 3 months
3. Eastern Cooperative Oncology Group (ECOG) performance status 0-2

Laboratory/Radiology

1. Adequate hepatic function, with serum ALT ≤ 3.5 times the upper limit of normal and serum direct bilirubin ≤ 2 mg/dL (34 µmol/L) within 14 days prior to randomization
2. Uric acid, if elevated, must be corrected to within laboratory normal range prior to dosing
3. Absolute neutrophil count (ANC) ≥ 1.0 × 109/L within 14 days prior to randomization independent of G-CSF for ≥ 1 week and pegylated G-CSF for ≥ 2 weeks
4. Hemoglobin ≥ 8 g/dL (80 g/L) within 14 days prior to randomization (subjects may be receiving red blood cell [RBC] transfusions in accordance with institutional guidelines)
5. Screening platelet count ≥ 50 × 109/L independent of platelet transfusions for at least 2 weeks
6. Creatinine clearance (CrCl) ≥ 15 mL/minute within 7 days prior to randomization, either measured or calculated using a standard formula (eg, Cockcroft and Gault)
7. LVEF ≥ 40% within 30 days before Cycle 1 Day 1. 2-D Transthoracic Echocardiogram (ECHO) is the preferred method of evaluation; MUGA is acceptable if ECHO is not available.

Exclusion Criteria:

Disease-related

1. Glucocorticoid therapy (prednisone > 10 mg/day or equivalent) within the last three weeks
2. POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
3. Chemotherapy with approved or investigative anticancer therapeutics including steroid therapy within the three weeks prior to first dose (unless enrolling on this study after progression CMAP compassionate use carfilzomib protocol, in which case subject may proceed with current study treatment on next expected date of treatment)
4. Radiation therapy or immunotherapy in the previous four weeks; localized radiation therapy within 1 week prior to first dose
5. Participation in an investigational therapeutic study within three weeks or within five drug half-lives (t1/2) prior to first dose, whichever time is greater (unless enrolling after progression on CMAP compassionate use carfilzomib protocol)

Concurrent Conditions

1. Pregnant or lactating females
2. Major surgery within 21 days prior to randomization
3. Acute active infection requiring treatment (systemic antibiotics, antivirals, or antifungals) within 14 days prior to randomization
4. Known human immunodeficiency virus infection
5. Known active hepatitis B or C infection
6. Unstable angina or myocardial infarction within 4 months prior to randomization, NYHA Class III or IV heart failure, uncontrolled angina, history of severe coronary artery disease, severe uncontrolled ventricular arrhythmias, sick sinus syndrome, or electrocardiographic evidence of acute ischemia or Grade 3 conduction system abnormalities unless subject has a pacemaker
7. Uncontrolled hypertension or uncontrolled diabetes within 14 days prior to randomization
8. Nonhematologic malignancy within the past 3 years with the exception of a) adequately treated basal cell carcinoma, squamous cell skin cancer, or thyroid cancer; b) carcinoma in situ of the cervix or breast; c) prostate cancer of Gleason Grade 6 or less with stable prostate-specific antigen levels; or d) cancer considered cured by surgical resection or unlikely to impact survival during the duration of the study, such as localized transitional cell carcinoma of the bladder or benign tumors of the adrenal or pancreas
9. Significant neuropathy (Grades 3-4, or Grade 2 with pain) within 14 days prior to randomization
10. Known history of allergy to Captisol® (a cyclodextrin derivative used to solubilize carfilzomib)
11. Contraindication to any of the required concomitant drugs or supportive treatments, including antiviral drugs, or intolerance to hydration due to preexisting pulmonary or cardiac impairment
12. Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis within 14 days prior to randomization
13. Any other clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-09; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajai Chari, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carfilzomib
Started | 13
Completed | 0
Not Completed | 13
Not completed — Adverse Event | 1
Not completed — Disease Progression | 12

BASELINE CHARACTERISTICS:
Arm/Group | Carfilzomib
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: years] | 62.9 [49 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Age >65 years [Count of Participants; unit: Participants] | 6
ECOG Performance Status [Count of Participants; unit: Participants] — The Eastern Cooperative Oncology Group (ECOG) measures level of functioning in terms of daily living abilities:
  0. - Fully active, able to carry on all pre-disease performance without restriction
  1. - Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. - Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  Participants
    0 | 5
    1 | 5
    2 | 3
ISS Staging [Count of Participants; unit: Participants] — The International Staging System (ISS): The ISS is based on the assessment of two blood test results: beta 2-microglobulin (ß2-M) and albumin.
  Stage I - ß2-M < 3.5 mg/dL and albumin =3.5 g/dL Stage II - Neither stage I nor stage III Stage III - ß2-M ≥ 5.5 mg/L
  Participants
    Stage 1 | 5
    Stage 2 | 5
    Stage 3 | 3
Immunoglobulin subtype [Count of Participants; unit: Participants]
  IgG | 10
  IgA | 3
  IgM | 0
  none | 0
Light-chain subtype [Count of Participants; unit: Participants]
  K | 7
  L | 6
FISH [Count of Participants; unit: Participants] — Fluorescence in situ hybridization (FISH), a molecular cytogenetic technique that tags genetic material with fluorescent molecules. FISH is useful for identifying chromosomes and parts of chromosomes, deciphering chromosome rearrangements, detecting chromosome abnormalities, and detecting and mapping genes.
  Participants
    Normal | 7
    Any abnormality | 6
Prior therapies since diagnosis [Median (Full Range); unit: years] | 7 [2 to 10]
Number of prior regimens [Median (Full Range); unit: prior regimens] | 5 [2 to 10]
Prior therapy [Number; unit: participants]
  Dexamethasone : Exposed | 13
  Dexamethasone : Refractory | 13
  Thalidomide : Exposed | 7
  Thalidomide : Refractory | 1
  Lenalidomide : Exposed | 13
  Lenalidomide : Refractory | 9
  Pomalidomide : Exposed | 8
  Pomalidomide : Refractory | 8
  Bortezomib : Exposed | 13
  Bortezomib : Refractory | 9
Prior Autologous Stem Cell Transplant [Count of Participants; unit: Participants] | 7
Carfilzomib Regimen Combination [Count of Participants; unit: Participants]
  Carfilzomib Regimen Combination | 13
  Weekly 40 mg DEX | 11
  Pomalidomide, DEX | 2
  Cyclophosphamide, DEX | 2
  Ibrutinib, DEX | 1
  Bendamustine | 1

OUTCOME MEASURES:

1. Primary Outcome: Safety and Efficacy of High Dose Carfilzomib
Description: The safety and efficacy of high dose carfilzomib who developed disease progression on the standard dosing and schedule of carfilzomib as measured by number of participants with adverse events
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 13
Participants
  Serious Adverse Events | 3
  Other than Serious Adverse Events | 13

2. Secondary Outcome: Progression Free Survival (PFS)
Time Frame: up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 12
months | 3.8 [1 to 12]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Overall Response Rate defined in categories
Time Frame: up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Carfilzomib
Number analyzed (Participants) | 12
Participants
  Complete Response | 0
  Very Good Partial Response | 1
  Partial Response | 4
  Minor Response | 2
  Stable Disease | 4

4. Secondary Outcome: Duration of Response to High Dose Carfilzomib
Time Frame: up to 4 years
Measure: Median (Full Range); unit: months
Arm/Group | Carfilzomib
Number analyzed (Participants) | 12
months | 9 [1 to 13]

5. Secondary Outcome: Markers of ER Stress
Description: The markers of ER stress signaling (both apoptotic and prosurvival) in MM cells from patients in this study and to determine if the balance of apoptotic versus prosurvival signaling changes upon recapture of response with carfilzomib dose escalation relative to the time of study entry.
Time Frame: up to 4 years
Population: data not collected
Arm/Group | Carfilzomib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Carfilzomib
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carfilzomib (N=13)
Acute Pulmonary Embolism (Blood and lymphatic system disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Carfilzomib (N=13)
Acute dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Acute renal failure (Renal and urinary disorders) | 1 (1)
alanine aminotransferase increased (Metabolism and nutrition disorders) | 1 (1)
alkaline phosphatase increased (Metabolism and nutrition disorders) | 1 (2)
anemia (Blood and lymphatic system disorders) | 8 (33)
ankle swelling (Metabolism and nutrition disorders) | 1 (1)
anorexia (General disorders) | 1 (1)
anterolisthesis of L5 over S1 (Musculoskeletal and connective tissue disorders) | 1 (1)
asparate aminotransferase increased (Metabolism and nutrition disorders) | 3 (3)
bilateral lower extremity leg pain (Musculoskeletal and connective tissue disorders) | 1 (2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
bilateral hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
cellulitis (Infections and infestations) | 1 (1)
chest heaviness (General disorders) | 1 (1)
chest pain (Respiratory, thoracic and mediastinal disorders) | 2 (4)
constipation (Gastrointestinal disorders) | 4 (4)
cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
creatinine elevated (Renal and urinary disorders) | 4 (4)
decreased creatinine clearance (Renal and urinary disorders) | 1 (1)
diaphoresis (General disorders) | 1 (1)
dizziness (General disorders) | 1 (1)
drift when walking (Nervous system disorders) | 1 (1)
dyspepsia (Gastrointestinal disorders) | 1 (1)
ejection fraction drop (Cardiac disorders) | 2 (2)
Elevated bilirubin (Metabolism and nutrition disorders) | 1 (1)
elevated GGT (Metabolism and nutrition disorders) | 1 (1)
epigastric pain (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 3 (4)
gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
hallucinations (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 6 (19)
high blood pressure (General disorders) | 1 (1)
hypercalcemia (Metabolism and nutrition disorders) | 6 (6)
hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
hypernatremia (Metabolism and nutrition disorders) | 1 (1)
hyperphostphatemia (Metabolism and nutrition disorders) | 3 (4)
hypertension (Cardiac disorders) | 7 (22)
hypertension chronic and intermittent fluctuation (Cardiac disorders) | 1 (1)
hypokalemia (Metabolism and nutrition disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
intermittent sternal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
lower extremity edema (Blood and lymphatic system disorders) | 1 (1)
left rib pain (Musculoskeletal and connective tissue disorders) | 1 (1)
left thigh pain (Musculoskeletal and connective tissue disorders) | 1 (1)
leukocyte count decreased (Blood and lymphatic system disorders) | 3 (3)
lymphocyte count decreased (Blood and lymphatic system disorders) | 3 (18)
lymphopenia (Blood and lymphatic system disorders) | 1 (1)
malaise (General disorders) | 1 (1)
minor cramps (Musculoskeletal and connective tissue disorders) | 1 (1)
nausea (General disorders) | 2 (5)
neuropathy (Nervous system disorders) | 1 (1)
neutrophil count decreased (Blood and lymphatic system disorders) | 4 (38)
non productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pain (General disorders) | 3 (3)
left mandible pain (General disorders) | 1 (1)
platelet count decreased (Blood and lymphatic system disorders) | 7 (29)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pruritic reddish hands with pain on hands wrist and arms (Skin and subcutaneous tissue disorders) | 1 (1)
right iliac bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
right rib pain (Musculoskeletal and connective tissue disorders) | 2 (3)
seizure (Nervous system disorders) | 1 (1)
shakiness/weakness (General disorders) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2)
sinusitis (General disorders) | 1 (1)
swelling in lower ankles (Blood and lymphatic system disorders) | 1 (1)
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (3)
vaginal pain (Reproductive system and breast disorders) | 1 (1)
vomiting (General disorders) | 1 (3)
weight loss (General disorders) | 1 (1)
wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
white blood cell decrease (Cardiac disorders) | 1 (1)
yeast infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes